CLINICAL TRIAL: NCT03800836
Title: A Phase Ib, Open-Label, Multicenter Study Evaluating the Safety and Efficacy of Ipatasertib in Combination With Atezolizumab and Paclitaxel or Nab-Paclitaxel in Patients With Locally Advanced or Metastatic Triple-Negative Breast Cancer
Brief Title: A Study to Evaluate the Safety and Efficacy of Ipatasertib in Combination With Atezolizumab and Paclitaxel or Nab-Paclitaxel in Participants With Locally Advanced or Metastatic Triple-Negative Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO40151; 2017-001957-15 (EudraCT Number)
Record Dates: First submitted 2019-01-07; First posted 2019-01-11 (Actual); Results first posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ipatasertib; Paclitaxel; atezolizumab; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (15):
- Arm A1: Ipat + Atezo + Pacl (Experimental): Safety Run-In (Cohort 1): Participants will receive ipatasertib orally daily on Days 1-21 of each 28 day cycle, and atezolizumab will be administered by intravenous (IV) infusion on Days 1 and 15 of each 28 day cycle. Paclitaxel will be administered by IV infusion on Days 1, 8, and 15 of each 28 day cycle. All participants in this cohort will continue to be treated until loss of clinical benefit, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Ipatasertib; Drug: Paclitaxel; Drug: Atezolizumab
- Arm A2: Ipat + Atezo + Pacl (Experimental): Expansion (Cohort 1): Participants will receive ipatasertib orally daily on Days 1-21 of each 28 day cycle, and atezolizumab will be administered by intravenous (IV) infusion on Days 1 and 15 of each 28 day cycle. Paclitaxel will be administered by IV infusion on Days 1, 8, and 15 of each 28 day cycle. All participants in this cohort will continue to be treated until loss of clinical benefit, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Ipatasertib; Drug: Paclitaxel; Drug: Atezolizumab
- Arm A3: Ipat + Atezo + Pacl (Experimental): Expansion (Cohort 1): Participants will receive ipatasertib orally daily on Days 1-21 of each 28 day cycle, and atezolizumab will be administered by intravenous (IV) infusion on Days 1 and 15 of each 28 day cycle. Paclitaxel will be administered by IV infusion on Days 1, 8, and 15 of each 28 day cycle. All participants in this cohort will continue to be treated until loss of clinical benefit, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Ipatasertib; Drug: Paclitaxel; Drug: Atezolizumab
- Arm B1: Ipat + Atezo + Nab-Pacl (Experimental): Safety Run-In (Cohort 1): Participants will receive ipatasertib orally daily on Days 1-21 of each 28 day cycle, and atezolizumab will be administered by IV infusion on Days 1 and 15 of each 28 day cycle. Nab-paclitaxel will be administered by IV infusion on Days 1, 8, and 15 of each 28 day cycle. All participants in this cohort will continue to be treated until loss of clinical benefit, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Ipatasertib; Drug: Atezolizumab; Drug: Nab-Paclitaxel
- Arm B2: Ipat + Atezo + Nab-Pacl (Experimental): Expansion (Cohort 1): Participants will receive ipatasertib orally daily on Days 1-21 of each 28 day cycle, and atezolizumab will be administered by IV infusion on Days 1 and 15 of each 28 day cycle. Nab-paclitaxel will be administered by IV infusion on Days 1, 8, and 15 of each 28 day cycle. All participants in this cohort will continue to be treated until loss of clinical benefit, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Ipatasertib; Drug: Atezolizumab; Drug: Nab-Paclitaxel
- Arm C1: (Ipat + Pacl) (2 weeks) + Atezo (Experimental): Safety Run-In (Cohort 1): Participants will receive a 2-week lead in of ipatasertib in combination with paclitaxel, followed by atezolizumab in an initial 28-day (1 cycle) period. Ipatasertib will be administered orally daily on Days 1-21, with paclitaxel administered by IV infusion on Days 1, 8 and 15. Atezolizumab will be administered by IV infusion on Day 15. In all subsequent treatment cycles, ipatasertib will be administered orally daily on Days 1-21, paclitaxel will be administered by IV infusion on Days 1, 8, and 15 and atezolizumab will be administered by IV infusion on Days 1 and 15. All participants in this cohort will continue to be treated until loss of clinical benefit, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Ipatasertib; Drug: Paclitaxel; Drug: Atezolizumab
- Arm C2 (Ipat + Pacl) (2 weeks) + Atezo (Experimental): Expansion (Cohort 1): Participants will receive a 2-week lead in of ipatasertib in combination with paclitaxel, followed by atezolizumab in an initial 28-day (1 cycle) period. Ipatasertib will be administered orally daily on Days 1-21, with paclitaxel administered by IV infusion on Days 1, 8 and 15. Atezolizumab will be administered by IV infusion on Day 15. In all subsequent treatment cycles, ipatasertib will be administered orally daily on Days 1-21, paclitaxel will be administered by IV infusion on Days 1, 8, and 15 and atezolizumab will be administered by IV infusion on Days 1 and 15. All participants in this cohort will continue to be treated until loss of clinical benefit, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Ipatasertib; Drug: Paclitaxel; Drug: Atezolizumab
- Arm D1: (Atezo + Pacl) (2 weeks) + Ipat (Experimental): Safety Run-In (Cohort 1): Participants will receive a 2-week lead in of atezolizumab in combination with paclitaxel, followed by ipatasertib in an initial 28-day (1 cycle) period. Atezolizumab will be administered via IV infusion on Days 1 and 15, with paclitaxel administered by IV infusion on Days 1, 8 and 15. Ipatasertib will be administered orally daily on Days 15-21. In all subsequent treatment cycles, ipatasertib will be administered orally daily on Days 1-21, paclitaxel will be administered by IV infusion on Days 1, 8, and 15 and atezolizumab will be administered by IV infusion on Days 1 and 15. All participants in this cohort will continue to be treated until loss of clinical benefit, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Ipatasertib; Drug: Paclitaxel; Drug: Atezolizumab
- Arm D2: (Atezo + Pacl) (2 weeks) + Ipat (Experimental): Expansion (Cohort 1): Participants will receive a 2-week lead in of atezolizumab in combination with paclitaxel, followed by ipatasertib in an initial 28-day (1 cycle) period. Atezolizumab will be administered via IV infusion on Days 1 and 15, with paclitaxel administered by IV infusion on Days 1, 8 and 15. Ipatasertib will be administered orally daily on Days 15-21. In all subsequent treatment cycles, ipatasertib will be administered orally daily on Days 1-21, paclitaxel will be administered by IV infusion on Days 1, 8, and 15 and atezolizumab will be administered by IV infusion on Days 1 and 15. All participants in this cohort will continue to be treated until loss of clinical benefit, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Ipatasertib; Drug: Paclitaxel; Drug: Atezolizumab
- Arm E: Ipat + Atezo (Experimental): Participants (Cohort 2) will receive Ipatasertib orally daily on Days 1-28 of Cycle 1 (35-day cycle) and on Days 1-21 of subsequent cycles (28-day cycles). Atezolizumab will be administered by IV infusion on Days 8 and 22 of Cycle 1 and on Days 1 and 15 of subsequent cycles. All participants in this cohort will continue to be treated until loss of clinical benefit, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Ipatasertib; Drug: Atezolizumab
- Arm F1: Ipat + Atezol + AC / Ipat + Atezo + Pacl (Experimental): Safety Run-In (Cohort 3): Participants will receive in Cycles 1 and 2 (28 day cycles), Ipatasertib orally daily on Days 1-21, Atezolizumab via IV infusion on Days 1 and 15 and AC (Doxorubicin and Cyclophosphamide) via IV infusion on Days 1 and 15. In Cycles 3-5, participants will receive Ipatasertib orally daily on Days 1-21, Atezolizumab via IV infusion on Days 1 and 15, with Paclitaxel administered by IV infusion on Days 1, 8, 15 and 22. All participants in this cohort will continue to be treated for five cycles (28-day cycles; 20 weeks) or until disease progression or unacceptable toxicity, whichever occurs first.
  Interventions: Drug: Ipatasertib; Drug: Paclitaxel; Drug: Atezolizumab; Drug: AC
- Arm F2: Ipat + Atezol + AC / Ipat + Atezo + Pacl (Experimental): Expansion (Cohort 3): Participants will receive in Cycles 1 and 2 (28 day cycles), Ipatasertib orally daily on Days 1-21, Atezolizumab via IV infusion on Days 1 and 15 and AC (Doxorubicin and Cyclophosphamide) via IV infusion on Days 1 and 15. In Cycles 3-5, participants will receive Ipatasertib orally daily on Days 1-21, Atezolizumab via IV infusion on Days 1 and 15, with Paclitaxel administered by IV infusion on Days 1, 8, 15 and 22. All participants in this cohort will continue to be treated for five cycles (28-day cycles; 20 weeks) or until disease progression or unacceptable toxicity, whichever occurs first.
  Interventions: Drug: Ipatasertib; Drug: Paclitaxel; Drug: Atezolizumab; Drug: AC
- Arm G1: Ipat + Atezol + AC / Ipat + Atezo + Pacl (Experimental): Safety Run-In (Cohort 3): Participants will receive in Cycles 1 and 2 (28 day cycles), Ipatasertib orally daily on Days 1-21, Atezolizumab via IV infusion on Days 1 and 15 and AC (Doxorubicin and Cyclophosphamide) via IV infusion on Days 1 and 15. In Cycles 3-5, participants will receive Ipatasertib orally daily on Days 1-21, Atezolizumab via IV infusion on Days 1 and 15, with Paclitaxel administered by IV infusion on Days 1, 8, 15 and 22. All participants in this cohort will continue to be treated for five cycles (28-day cycles; 20 weeks) or until disease progression or unacceptable toxicity, whichever occurs first.
  Interventions: Drug: Ipatasertib; Drug: Paclitaxel; Drug: Atezolizumab; Drug: AC
- Arm G2: Ipat + Atezol + AC / Ipat + Atezo + Pacl (Experimental): Expansion (Cohort 3): Participants will receive in Cycles 1 and 2 (28 day cycles), Ipatasertib orally daily on Days 1-21, Atezolizumab via IV infusion on Days 1 and 15 and AC (Doxorubicin and Cyclophosphamide) via IV infusion on Days 1 and 15. In Cycles 3-5, participants will receive Ipatasertib orally daily on Days 1-21, Atezolizumab via IV infusion on Days 1 and 15, with Paclitaxel administered by IV infusion on Days 1, 8, 15 and 22. All participants in this cohort will continue to be treated for five cycles (28-day cycles; 20 weeks) or until disease progression or unacceptable toxicity, whichever occurs first.
  Interventions: Drug: Ipatasertib; Drug: Paclitaxel; Drug: Atezolizumab; Drug: AC
- Arm H: Ipat + Atezo + Pacl (Experimental): Participants (Cohort 4) will receive ipatasertib orally daily on Days 1-21 of each 28 day cycle, and atezolizumab will be administered by intravenous (IV) infusion on Days 1 and 15 of each 28 day cycle. Paclitaxel will be administered by IV infusion on Days 1, 8, and 15 of each 28 day cycle. All participants in this cohort will continue to be treated until loss of clinical benefit, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Ipatasertib; Drug: Paclitaxel; Drug: Atezolizumab

INTERVENTIONS:
Drug: Ipatasertib — Ipatasertib will be administered at a dose of 400 milligrams (mg) orally daily on Days 1-21 of each 28 day cycle for all arms except for arms F1/F2 where it will be administered at a dose of 300 milligrams (mg) orally daily for the first two cycles and 400 mg for the remaining three cycles.
Drug: Paclitaxel — Paclitaxel will be administered at a dose of 80 milligrams per square meter (mg/m^2) as IV infusion on Days 1, 8, and 15 of each 28 day cycle for all arms, with the exceptions of Arms F1, F2, G1 and G2, where it will be also administered on Day 22 as well, of each 28 day cycle.
  Arms: Arm A1: Ipat + Atezo + Pacl; Arm A2: Ipat + Atezo + Pacl; Arm A3: Ipat + Atezo + Pacl; Arm C1: (Ipat + Pacl) (2 weeks) + Atezo; Arm C2 (Ipat + Pacl) (2 weeks) + Atezo; Arm D1: (Atezo + Pacl) (2 weeks) + Ipat; Arm D2: (Atezo + Pacl) (2 weeks) + Ipat; Arm F1: Ipat + Atezol + AC / Ipat + Atezo + Pacl; Arm F2: Ipat + Atezol + AC / Ipat + Atezo + Pacl; Arm G1: Ipat + Atezol + AC / Ipat + Atezo + Pacl; Arm G2: Ipat + Atezol + AC / Ipat + Atezo + Pacl; Arm H: Ipat + Atezo + Pacl
Drug: Atezolizumab — Atezolizumab will be administered by IV infusion at a fixed dose of 840 mg on Days 1 and 15 of each 28 day cycle for all arms, although in Arms C1/C2, it will be administered on Day 15 of Cycle 1 followed by Days 1 and 15 in subsequent cycles.
Drug: Nab-Paclitaxel — Nab-paclitaxel will be administered by IV infusion at a dose of 100 mg/m^2 on Days 1, 8, and 15 of each 28 day cycle.
  Arms: Arm B1: Ipat + Atezo + Nab-Pacl; Arm B2: Ipat + Atezo + Nab-Pacl
Drug: AC — AC (Doxorubicin and Cyclophosphamide) will be administered by IV infusion at 60 mg/m^2 and 600 mg/m^2 respectively on Days 1 and 15 of Cycles 1 and 2 for Arms F1, F2, G1 and G2.
  Arms: Arm F1: Ipat + Atezol + AC / Ipat + Atezo + Pacl; Arm F2: Ipat + Atezol + AC / Ipat + Atezo + Pacl; Arm G1: Ipat + Atezol + AC / Ipat + Atezo + Pacl; Arm G2: Ipat + Atezol + AC / Ipat + Atezo + Pacl

SUMMARY:
This is a study consisting of four cohorts in this setting. In Cohort 1, the safety and efficacy of ipatasertib (ipat) in combination with atezolizumab (atezo) and paclitaxel (pac) or nab-paclitaxel will be evaluated for participants with locally advanced or metastatic triple-negative breast cancer (TNBC) who have not previously received chemotherapy. In Cohort 2, ipatasertib and atezolizumab (with no chemotherapy), will be administered to participants with locally advanced or metastatic TNBC. In Cohort 3, the safety and efficacy of neoadjuvant ipatasertib, atezolizumab, doxorubicin and cyclophosphamide (AC) (Ipat + Atezo + AC) followed by Ipat + Atezo + Pac will be evaluated in participants with locally advanced Type 2-4 (T2-4) TNBC. In Cohort 4, the safety and efficacy of Ipat + Atezo + Pac will be evaluated in participants with PD-L1 (Programmed Death-Ligand-1) positive locally advanced or metastatic TNBC that is not amenable to resection and who have not previously received chemotherapy in the advanced setting.

ELIGIBILITY:
Inclusion Criteria:

General:

* Eastern Cooperative Oncology Group Performance Status of 0 or 1.
* Adequate hematologic and organ function.
* For Cohorts 1, 2 and 4: Life expectancy of at least 6 months.
* For men and women of child bearing potential: agreement to remain abstinent or use protocol defined contraceptive measures during the treatment period and for at least 28 days after the last dose of ipatasertib, 6 months after the last dose of paclitaxel, nab-paclitaxel, or doxorubicin, and 12 months after the last dose of cyclophosphamide, and 5 months after the last dose of atezolizumab, whichever occurs later along with refraining from donating sperm or eggs during this same period.

Disease-specific:

* For Cohorts 1, 2 and 4: histologically documented TNBC that is locally advanced or metastatic and is not amenable to resection with curative intent.
* For Cohort 2: disease progression following one or two lines of systemic therapy for inoperable locally advanced or metastatic TNBC.
* For Cohorts 1, 2 and 4: measurable disease according to RECIST v1.1 criteria.
* For Cohort 2: Treated brain or spinal cord metastases are allowed if participants have stable disease and are not on steroid treatment.
* For Cohort 3: histologically documented TNBC with a primary breast tumour size of > 2 cm by at least one radiographic or clinical measurement and disease stage at presentation of cT2-4 cN0-3 cM0.
* For Cohort 3: participant agreement to undergo appropriate surgical management, including axillary lymph node surgery and partial or total mastectomy, after completion of neoadjuvant treatment.
* For Cohort 4: participants must have centrally confirmed PD-L1-positive tumour.

Exclusion Criteria:

General:

* History of malabsorption syndrome or other condition that would interfere with enteral absorption or results in the inability or unwillingness to swallow pills.
* Active infection requiring antibiotics.
* History of or current evidence of HIV infection.
* Known clinically significant history of liver disease.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 of Cycle 1 or anticipation of need for a major surgical procedure (other than anticipated breast surgery for Cohort 3) during the course of the study.
* Pregnant or breastfeeding.
* New York Heart Association (NYHA) Class II, III, or IV heart failure; left ventricular ejection fraction < 50%; or active ventricular arrhythmia requiring medication.
* Treatment with approved or investigational cancer therapy within 14 days prior to Day 1 of Cycle 1.
* Prior treatment with an Akt inhibitor.

Disease-specific:

* For Cohorts 1 and 4: history of or known presence of brain or spinal cord metastases.
* For Cohorts 1 and 4: participants who have received previous systemic therapy for inoperable locally advanced or metastatic TNBC, including chemotherapy, immune checkpoint inhibitors, or targeted agents.
* Unresolved, clinically significant toxicity from prior therapy, except for alopecia and Grade 1 peripheral neuropathy.
* Participants who have received palliative radiation treatment to peripheral sites (e.g., bone metastases) for pain control and whose last treatment was completed 14 days prior to Day 1 of Cycle 1 and have recovered from all acute, reversible effects.
* Uncontrolled pleural effusion, pericardial effusion, or ascites.
* Uncontrolled tumor related complications.
* Uncontrolled hypercalcaemia or symptomatic hypercalcaemia requiring continued use of bisphosphonate therapy.
* Malignancies other than breast cancer within 5 years prior to Day 1 of Cycle 1.
* For Cohort 3, participants with the following are excluded: [1] prior history of invasive breast cancer; [2] prior systemic therapy for treatment and/or prevention of invasive breast cancer; [3] previous therapy with anthracyclines or taxanes for any malignancy; [4] bilateral breast cancer; [5] undergone incisional and/or excisional biopsy of primary tumor and/or axillary lymph nodes; [6] undergone axillary lymph node dissection (ALND) prior to initiation of neoadjuvant therapy; [6] history of other malignancy within 5 years prior to screening; [7] history of cerebrovascular accident within 12 months prior to initiation of study treatment; [8] cardiopulmonary dysfunction; [9] known allergy or hypersensitivity to the components of cyclophosphamide/doxorubicin formulations and filgrastim or pegfilgrastim formulations; [10] severe infection within 4 weeks prior to initiation of study treatment; [11] treatment with therapeutic oral or IV (Intravenous) antibiotics within 2 weeks prior to initiation of study treatment and [12] prior treatment with CD137 agonists or immune checkpoint - blockade therapies.

Ipatasertib-specific:

* History of Type I or Type II diabetes mellitus requiring insulin.
* Grade >= 2 uncontrolled or untreated hypercholesterolemia or hypertriglyceridemia.
* History of or active inflammatory bowel disease or active bowel inflammation.
* Clinically significant lung disease.
* Treatment with strong CYP3A inhibitors or strong CYP3A inducers.

Atezolizumab-specific:

* Active or history of autoimmune disease or immune deficiency.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan.
* Prior allogeneic stem cell or solid organ transplantation.
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during treatment with atezolizumab or within 5 months after the last dose of atezolizumab.
* History of hypersensitivity reactions to study drug or any component of the study drug formulation.
* Treatment with systemic immunostimulatory agents and immunosuppressive medication treatment, or anticipation of need for systemic immunosuppressive medication during the course of the study.

Paclitaxel-specific:

- Grade >= 2 peripheral neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (18):
- Pacific Shores Medical Group, Long Beach, California, United States
- Australia (3):
  - St Vincents Hospital; Cardiopulmonary transplant Ambulatory Care Dept, Darlinghurst, New South Wales
  - Austin Hospital, Heidelberg, Victoria
  - Peter MacCallum Cancer Center, North Melbourne, Victoria
- France (5):
  - Institut de Cancerologie de l Ouest, Angers
  - Institut Bergonie, Bordeaux
  - Centre Georges Francois Leclerc, Dijon
  - Institut Curie, Paris
  - Gustave Roussy, Villejuif
- Spain (7):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Clinico San Carlos; Servicio de Oncologia, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz., Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Centro Integral Oncologico Clara Campal (CIOCC); Dirección Médica, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
- United Kingdom (2):
  - Barts Cancer Institute, London
  - Nottingham University Hospitals NHS Trust, Nottingham

REFERENCES:
- [Derived] Schmid P, Turner NC, Barrios CH, Isakoff SJ, Kim SB, Sablin MP, Saji S, Savas P, Vidal GA, Oliveira M, O'Shaughnessy J, Italiano A, Espinosa E, Boni V, White S, Rojas B, Freitas-Junior R, Chae Y, Bondarenko I, Lee J, Torres Mattos C, Martinez Rodriguez JL, Lam LH, Jones S, Reilly SJ, Huang X, Shah K, Dent R. First-Line Ipatasertib, Atezolizumab, and Taxane Triplet for Metastatic Triple-Negative Breast Cancer: Clinical and Biomarker Results. Clin Cancer Res. 2024 Feb 16;30(4):767-778. doi: 10.1158/1078-0432.CCR-23-2084. PMID 38060199

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in this study from 13 February 2018 to 16 March 2022.
Pre-assignment Details: 139 participants were enrolled, 2 were not treated and excluded from analyses. 137 participants were enrolled in either Cohort 1 (Arms A [A1,2,3], B [B1,2], C [C1,2], and D [D1,2]), Cohort 2 (Arm E) or Arm F1 in Cohort 3. Sponsor made decision not to continue study enrollment before arms F2, G1, G2 (Cohort 3) and H (Cohort 4) enrolled any participants.
Groups:
- Cohort 1-Arm A: Participants with locally advanced or metastatic triple-negative breast cancer (TNBC) who had not previously received chemotherapy in the advanced setting received 400 milligrams (mg) of ipatasertib (Ipat) orally, once daily (QD) on Days 1-21, 840 mg intravenous (IV) of atezolizumab (Atezo) on Days 1 and 15, and 80 milligrams per square meter (mg/m^2) IV paclitaxel (Pac) on Days 1, 8, and 15 of each 28-day cycle. Following completion of a safety run-in cohort (A1), subsequent expansion arms enrolled (A2 and A3). All participants in Arm A continued to receive treatment until loss of clinical benefit, unacceptable toxicity, withdrawal of consent, or end of the study.
- Cohort 1-Arm B: Participants with locally advanced or metastatic TNBC who had not previously received chemotherapy in the advanced setting received 400 mg of Ipat orally, QD on Days 1-21, 840 mg IV of Atezo on Days 1 and 15, and 100 mg/m^2 IV nab-paclitaxel (Nab-Pac) on Days 1, 8, and 15 of each 28-day cycle. Following completion of a safety run-in cohort (B1), a subsequent expansion arm enrolled (B2). All participants in Arm B continued to receive treatment until loss of clinical benefit, unacceptable toxicity, withdrawal of consent, or end of the study.
- Cohort 1-Arm C: Participants with locally advanced or metastatic TNBC who had not previously received chemotherapy in the advanced setting received 400 mg of Ipat orally, QD on Days 1-21, 80 mg/m2 IV Pac on Days 1, 8, and 15 and 840 mg IV Atezo on Day 15 of Cycle 1 (28 day cycle). In Cycles ≥ 2, participants received 400 mg Ipat orally on Days 1-21, 840 mg IV Atezo on Days 1 and 15 and 80 mg/m2 IV Pac on Days 1, 8, and 15 of each 28-day Cycle. Following completion of the safety run-in cohort (C1), a subsequent expansion cohort (C2) enrolled. All participants in Arm C continued to receive treatment until loss of clinical benefit, unacceptable toxicity, withdrawal of consent, or end of the study.
- Cohort 1-Arm D: Participants with locally advanced or metastatic TNBC who had not previously received chemotherapy in the advanced setting received 840 mg IV Atezo on Days 1 and 15, 80 mg/m2 IV Pac on Days 1, 8, and 15 and 400 mg Ipat orally on days 15-21 of Cycle 1 (28 day cycle). In Cycles ≥ 2, participants received 400 mg Ipat orally on Days 1-21, 80 mg/m2 IV Pac on Days 1, 8, and 15 and 840 mg IV Atezo on Days 1 and 15 of each 28 day Cycle. Following completion of the safety run-in cohort (D1), a subsequent expansion cohort (D2) enrolled. All participants in Arm D continued to receive treatment until loss of clinical benefit, unacceptable toxicity, withdrawal of consent, or end of the study.
- Cohort 2-Arm E: Participants in the second-line and third-line setting with locally advanced or metastatic TNBC received 400 mg Ipat orally QD on Days 1-28 and 840 mg IV Atezo on Days 8 and 22 of Cycle 1 (Cycle 1 = 35 days). In Cycles ≥ 2, participants received 400 mg Ipat orally on Days 1-21 and 840 mg IV Atezo on Days 1 and 15 of each cycle (Cycles ≥ 2 = 28-days) until loss of clinical benefit, unacceptable toxicity, withdrawal of consent, or end of the study.
- Cohort 3-Arm F: Participants in the safety run-in stage (arm F1) with locally advanced T2-4 TNBC received 300 mg Ipat orally QD on Days 1-21, 840mg IV Atezo on Days 1 and 15, 60 mg/m2 IV doxorubicin and 600 mg/m2 IV cyclophosphamide on Days 1 and 15 of Cycles 1 and 2 (1 Cycle=28-days). Participants then received 400 mg Ipat orally QD on Days 1-21, 840mg IV Atezo on Days 1 and 15 and 80 mg/m2 IV Pac on Days 1, 8, 15, and 22 of Cycles 3-5, until completion of 5 cycles or disease progression or unacceptable toxicity, whichever occurred first.
Period: Overall Study
Arm/Group | Cohort 1-Arm A | Cohort 1-Arm B | Cohort 1-Arm C | Cohort 1-Arm D | Cohort 2-Arm E | Cohort 3-Arm F
Started | 71 | 20 | 13 | 12 | 17 | 6
Safety Population (Safety population included all participants who received any study treatment.) | 70 | 20 | 12 | 12 | 17 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 71 | 20 | 13 | 12 | 17 | 6
Not completed — Other | 2 | 1 | 0 | 2 | 0 | 1
Not completed — Lost to Follow-up | 2 | 0 | 1 | 1 | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 31 | 3 | 6 | 4 | 4 | 5
Not completed — Death | 34 | 16 | 5 | 5 | 10 | 0
Not completed — Symptomatic Deterioration | 1 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received any study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1-Arm A | Cohort 1-Arm B | Cohort 1-Arm C | Cohort 1-Arm D | Cohort 2-Arm E | Cohort 3-Arm F | Total
Number analyzed (Participants) | 70 | 20 | 12 | 12 | 17 | 6 | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (13.0) | 50.2 (9.6) | 46.4 (14.0) | 48.8 (9.6) | 52.1 (11.2) | 53.2 (7.4) | 53.4 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 20 | 12 | 12 | 17 | 6 | 137
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 5 | 0 | 0 | 1 | 0 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 1
  White | 55 | 15 | 11 | 9 | 17 | 6 | 113
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 8 | 5 | 1 | 2 | 0 | 0 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 3 | 1 | 0 | 5 | 2 | 18
  Not Hispanic or Latino | 51 | 14 | 9 | 11 | 11 | 4 | 100
  Not Stated | 7 | 2 | 2 | 0 | 1 | 0 | 12
  Unknown | 5 | 1 | 0 | 1 | 0 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1 and Cohort 4: Percentage of Participants With Objective Response (OR) as Assessed by Investigator Based on Response Evaluation Criteria in Solid Tumors (RECIST), Version (v) 1.1
Description: Objective Response Rate: percentage participants with confirmed complete response (CR) or partial response (PR) on 2 consecutive occasions >or= 4 weeks apart, as determined by investigator according to RECIST v1.1. CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR: at least a 30% decrease in sum of diameters of target lesions, taking as reference baseline sum diameters. Percentages have been rounded off. No participants were enrolled in cohort 4, hence no data reported.
Time Frame: From screening up to approximately 43.6 months
Population: Efficacy evaluable population included all enrolled participants who received at least one dose of study treatment, regardless of treatment allocation. Participants without a postbaseline tumor assessment were considered as non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1-Arm A | Cohort 1-Arm B | Cohort 1-Arm C | Cohort 1-Arm D
Number analyzed (Participants) | 70 | 20 | 12 | 12
percentage of participants | 51.4 [39.17 to 63.56] | 65.0 [40.78 to 84.61] | 66.7 [34.89 to 90.08] | 33.3 [9.92 to 65.11]

2. Secondary Outcome: Cohort 1 and Cohort 4: Duration of Response (DOR), as Determined by the Investigator According to RECIST v1.1
Description: DOR was defined as the time from the first occurrence of a documented confirmed CR or PR to the first date of recorded disease progression (PD), as determined by the investigator according to RECIST v1.1 or death from any cause. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduced in short axis to < 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. PD was defined as at least a 20% increase in the sum of diameter of target lesions, taking as reference the smallest sum on study (nadir) including baseline; the appearance of one or more new lesions. No participants were enrolled in cohort 4, and hence no data was reported. Participants who did not progress or died at time of analysis were censored at last disease assessment date.
Time Frame: From the date of first documented confirmed response (CR or PR) to disease progression or death due to any cause (up to approximately 43.6 months)
Population: Efficacy evaluable population included all enrolled participants who received at least one dose of study treatment, regardless of treatment allocation. Number analyzed are participants who had OR (i.e., a confirmed CR or PR).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1-Arm A | Cohort 1-Arm B | Cohort 1-Arm C | Cohort 1-Arm D
Number analyzed (Participants) | 36 | 13 | 8 | 4
months | 7.8 [5.6 to 12.9] | 7.3 [5.0 to 9.2] | 9.2 [3.9 to 14.7] | 4.8 [3.7 to NA] — The median and upper limit of confidence interval (CI) were not estimable due to less number of participants with events.

3. Primary Outcome: Cohort 3: Pathological Complete Response (pCR) Rate
Description: pCR rate was defined as the percentage of participants who had no residual invasive disease in the breast and no residual disease in the lymph nodes (ypT0/Tis ypN0 in the current American Joint Committee on Cancer (AJCC )staging system) based on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant therapy.
Time Frame: 2-6 weeks following last dose of study treatment (up to 69 weeks)
Population: Efficacy evaluable population included all enrolled participants who received at least one dose of study treatment, regardless of treatment allocation.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 3-Arm F
Number analyzed (Participants) | 6
percentage of participants | 50

4. Primary Outcome: Cohort 1, Cohort 2, Cohort 3 and Cohort 4: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any new disease or worsening of an existing disease are also considered as AEs. AEs were reported based on the National Cancer Institute Common Terminology Criteria for AEs, version 4.0 (NCI-CTCAE, v4.0). No participants were enrolled in cohort 3 Arm G and 4, and hence no data was reported.
Time Frame: Up until 90 days after the last dose of study treatment or until initiation of new systemic anti-cancer therapy, whichever occurs first (up to 4 years 1 month)
Population: Safety population included all participants who received any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1-Arm A | Cohort 1-Arm B | Cohort 1-Arm C | Cohort 1-Arm D | Cohort 2-Arm E | Cohort 3-Arm F
Number analyzed (Participants) | 70 | 20 | 12 | 12 | 17 | 6
Participants | 70 | 20 | 12 | 12 | 17 | 6

5. Secondary Outcome: Cohort 1 and Cohort 4: Progression-Free Survival (PFS), as Assessed by Investigator Based on RECIST v1.1
Description: PFS: time from enrollment to date of 1st recorded occurrence of PD, as determined by investigator according to RECIST v1.1 or death from any cause, whichever occurs first. PD: at least a 20% increase in sum of diameters of target lesions, taking as reference smallest sum on study (nadir) including baseline; appearance of one or more new lesions. Data for participants who did not experience PD or death was censored at last date of evaluable tumor assessment. No participants were enrolled in cohort 4, and hence no data was reported.
Time Frame: From enrollment up to disease progression or death due to any cause whichever occurs first (up to approximately 43.6 months)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1-Arm A | Cohort 1-Arm B | Cohort 1-Arm C | Cohort 1-Arm D
Number analyzed (Participants) | 70 | 20 | 12 | 12
months | 7.2 [5.3 to 7.4] | 6.6 [3.4 to 9.2] | 8.8 [5.6 to 12.9] | 6.5 [5.2 to 11.3]

6. Secondary Outcome: Cohort 1 and Cohort 4: Overall Survival (OS)
Description: OS was defined as the time from enrollment to death from any cause.
Time Frame: From enrollment up to death due to any cause (up to approximately 43.6 months).
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1-Arm A | Cohort 1-Arm B | Cohort 1-Arm C | Cohort 1-Arm D
Number analyzed (Participants) | 70 | 20 | 12 | 12
months | 28.3 [17.2 to 43.0] | 20.1 [11.1 to 30.8] | NA [21.2 to NA] — The median and upper limit of confidence interval (CI) were not estimable due to less number of participants with events. | NA [11.7 to NA] — The median and upper limit of CI were not estimable due to less number of participants with events.

7. Secondary Outcome: Cohort 1 and Cohort 4: Plasma Concentration of Ipatasertib
Description: Since, Cohort 4 did not enroll any participants, data is only reported for Cohort 1.
Time Frame: Day 15 Cycle 1: pre-dose and 1, 2, 4 and 6 hours post-dose, Day 15 Cycle2: predose and 1, 2, 4 and 6 hours post-dose and Day 15 Cycle 3 - post dose up to - 3 hours (each cycle is of 28 days)
Population: Pharmacokinetic (PK) evaluable population included all participants who had at least 1 evaluable PK concentration post ipatasertib administration. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at a given time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- Cohort 1- Arm A1: Participants with locally advanced or metastatic TNBC who had not previously received chemotherapy in the advanced setting received 400 mg of Ipat orally, QD on Days 1-21, 840 mg IV of Atezo on Days 1 and 15, and 80 mg/m^2 IV Pac on Days 1, 8, and 15 of each 28-day cycle during the safety run-in stage (A1) until loss of clinical benefit, unacceptable toxicity, withdrawal of consent, or end of the study.
- Cohort 1- A2: Participants with locally advanced or metastatic TNBC who had not previously received chemotherapy in the advanced setting received 400 mg of Ipat orally, QD on Days 1-21, 840 mg IV of Atezo on Days 1 and 15, and 80 mg/m^2 IV Pac on Days 1, 8, and 15 of each 28-day cycle in expansion stage A2 until loss of clinical benefit, unacceptable toxicity, withdrawal of consent, or end of the study.
- Cohort1- Arm A3: Participants with locally advanced or metastatic TNBC who had not previously received chemotherapy in the advanced setting received 400 mg of Ipat orally, QD on Days 1-21, 840 mg IV of Atezo on Days 1 and 15, and 80 mg/m^2 IV Pac on Days 1, 8, and 15 of each 28-day cycle in expansion stage A3 until loss of clinical benefit, unacceptable toxicity, withdrawal of consent, or end of the study.
- Cohort 1- Arm B1: Participants with locally advanced or metastatic TNBC who had not previously received chemotherapy in the advanced setting received 400 mg of Ipat orally, QD on Days 1-21, 840 mg IV of Atezo on Days 1 and 15, and 100 mg/m^2 IV Nab-Pac on Days 1, 8, and 15 of each 28-day cycle during the safety run-in stage (B1) until loss of clinical benefit, unacceptable toxicity, withdrawal of consent, or end of the study.
- Cohort 1- Arm B2: Participants with locally advanced or metastatic TNBC who had not previously received chemotherapy in the advanced setting received 400 mg of Ipat orally, QD on Days 1-21, 840 mg IV of Atezo on Days 1 and 15, and 100 mg/m^2 IV Nab-Pac on Days 1, 8, and 15 of each 28-day cycle in the expansion stage B2 until loss of clinical benefit, unacceptable toxicity, withdrawal of consent, or end of the study.
- Cohort 1- Arm C1: Participants with locally advanced or metastatic TNBC who had not previously received chemotherapy in the advanced setting received 400 mg of Ipat orally, QD on Days 1-21, 80 mg/m2 IV Pac on Days 1, 8, and 15 of Cycle 1 and 840 mg IV Atezo on Day 15 of Cycle 1 (1 Cycle=28days). In Cycles ≥ 2, participants received 400 mg Ipat orally on Days 1-21, 840 mg IV Atezo on Days 1 and 15 and 80 mg/m2 IV Pac on Days 1, 8, and 15 of each 28-day cycle during the safety run-in stage (C1) until loss of clinical benefit, unacceptable toxicity, withdrawal of consent, or end of the study.
- Cohort 1- Arm C2: Participants with locally advanced or metastatic TNBC who had not previously received chemotherapy in the advanced setting received 400 mg of Ipat orally, QD on Days 1-21, 80 mg/m2 IV Pac on Days 1, 8, and 15 of Cycle 1 and 840 mg IV Atezo on Day 15 of Cycle 1 (1Cycle=28days). In Cycles ≥ 2, participants received 400 mg Ipat orally on Days 1-21, 840 mg IV Atezo on Days 1 and 15 and 80 mg/m2 IV Pac on Days 1, 8, and 15 of each 28-day cycle in the expansion stage C2 until loss of clinical benefit, unacceptable toxicity, withdrawal of consent, or end of the study.
- Cohort 1- Arm D1: Participants with locally advanced or metastatic TNBC received 840 mg IV Atezo on Days 1 and 15, 80 mg/m2 IV Pac on Days 1, 8, and 15 and 400 mg Ipat orally on days 15-21 of Cycle 1. In Cycles ≥ 2, participants received 400 mg Ipat orally on Days 1-21, 80 mg/m2 IV Pac on Days 1, 8, and 15 and 840 mg IV Atezo on Days 1 and 15 of each 28-day Cycle during the safety run-in stage (D1) until loss of clinical benefit, unacceptable toxicity, withdrawal of consent, or end of the study.
- Cohort 1- Arm D2: Participants with locally advanced or metastatic TNBC received 840 mg IV Atezo on Days 1 and 15, 80 mg/m2 IV Pac on Days 1, 8, and 15 and 400 mg Ipat on days 15-21 of cycle 1. In Cycles ≥ 2, participants received 400 mg Ipat orally on Days 1-21, 80 mg/m2 IV Pac on Days 1, 8, and 15 and 840 mg IV Atezo on days 1 and 15 of each 28-day cycle in the expansion stage D2 until loss of clinical benefit, unacceptable toxicity, withdrawal of consent, or end of the study.
Arm/Group | Cohort 1- Arm A1 | Cohort 1- A2 | Cohort1- Arm A3 | Cohort 1- Arm B1 | Cohort 1- Arm B2 | Cohort 1- Arm C1 | Cohort 1- Arm C2 | Cohort 1- Arm D1 | Cohort 1- Arm D2
Number analyzed (Participants) | 6 | 14 | 50 | 6 | 14 | 6 | 6 | 6 | 6
nanograms per milliliter (ng/mL)
  Cycle 1 Day 15 Pre-dose: number analyzed (Participants) | 5 | 11 | 26 | 5 | 11 | 4 | 6 | 0 | 0
  Cycle 1 Day 15 Pre-dose | 47.9 (47.2) | 13.6 (783.4) | 29.4 (163.1) | 30.2 (37.1) | 46.9 (172.8) | 61.1 (94.3) | 77.3 (207.0) |  |
  Cycle 1 Day 15 1 hour Post-dose: number analyzed (Participants) | 5 | 10 | 25 | 5 | 10 | 0 | 0 | 0 | 0
  Cycle 1 Day 15 1 hour Post-dose | 507 (43.6) | 182 (167.0) | 258 (127.2) | 253 (128.0) | 219 (186.6) |  |  |  |
  Cycle 1 Day 15 2 hour Post-dose: number analyzed (Participants) | 5 | 10 | 33 | 5 | 10 | 0 | 0 | 6 | 5
  Cycle 1 Day 15 2 hour Post-dose | 318 (21.4) | 318 (47.8) | 421 (51.5) | 287 (35.7) | 282 (235.6) |  |  | 225 (41.9) | 190 (484.7)
  Cycle 1 Day 15 4 hour Post-dose: number analyzed (Participants) | 3 | 10 | 33 | 5 | 10 | 0 | 0 | 0 | 0
  Cycle 1 Day 15 4 hour Post-dose | 226 (32.7) | 255 (39.7) | 305 (40.8) | 225 (10.0) | 266 (78.1) |  |  |  |
  Cycle 1 Day 15 6 hour Post-dose: number analyzed (Participants) | 0 | 9 | 33 | 5 | 10 | 0 | 0 | 0 | 0
  Cycle 1 Day 15 6 hour Post-dose |  | 182 (39.2) | 233 (46.7) | 165 (25.0) | 186 (80.3) |  |  |  |
  Cycle 2 Day 15 Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 4 | 2
  Cycle 2 Day 15 Pre-dose |  |  |  |  |  | 44.9 (43.3) | 50.3 (31.4) | 29.2 (59.5) | 31.6 (53.1)
  Cycle 2 Day 15 1 hour Post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 4 | 2
  Cycle 2 Day 15 1 hour Post-dose |  |  |  |  |  | 260 (21.6) | 614 (34.2) | 232 (150.0) | 364 (81.4)
  Cycle 2 Day 15 2 hour Post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 4 | 2
  Cycle 2 Day 15 2 hour Post-dose |  |  |  |  |  | 575 (22.5) | 500 (18.3) | 311 (67.5) | 610 (36.7)
  Cycle 2 Day 15 4 hour Post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 3 | 2
  Cycle 2 Day 15 4 hour Post-dose |  |  |  |  |  | 402 (44.9) | 340 (29.9) | 258 (20.6) | 433 (41.7)
  Cycle 2 Day 15 6 hour Post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 5 | 3 | 2
  Cycle 2 Day 15 6 hour Post-dose |  |  |  |  |  | 253 (31.7) | 273 (15.3) | 162 (8.2) | 234 (32.6)
  Cycle 3 Day 15 1 to 3 hour Post-dose: number analyzed (Participants) | 0 | 11 | 26 | 4 | 9 | 6 | 5 | 6 | 4
  Cycle 3 Day 15 1 to 3 hour Post-dose |  | 126 (241.7) | 196 (133.7) | 134 (82.8) | 214 (130.8) | 127 (369.0) | 155 (282.3) | 233 (120.9) | 382 (87.9)

8. Secondary Outcome: Cohort 1 and Cohort 4: Plasma Concentration of Ipatasertib Metabolite M1 (G-037720)
Description: Since, Cohort 4 did not enroll any participants, data is only reported for Cohort 1.
Time Frame: Day 15 Cycle 1 - pre-dose and 1 hour, 2 hours, 4 hours and 6 hours post-dose, Day 15 Cycle2: predose and 1 hour, 2 hours, 4 hours and 6 hours post-dose and Day 15 Cycle 3 - post dose up to - 3 hours (each cycle is of 28 days)
Population: PK evaluable population included all participants who had at least 1 evaluable PK concentration post ipatasertib administration. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at a given time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Cohort 1-Arm A2: Participants with locally advanced or metastatic TNBC who had not previously received chemotherapy in the advanced setting received 400 mg of Ipat orally, QD on Days 1-21, 840 mg IV of Atezo on Days 1 and 15, and 80 mg/m^2 IV Pac on Days 1, 8, and 15 of each 28-day cycle in expansion stage A2 until loss of clinical benefit, unacceptable toxicity, withdrawal of consent, or end of the study.
- Cohort 1-Arm A3: Participants with locally advanced or metastatic TNBC who had not previously received chemotherapy in the advanced setting received 400 mg of Ipat orally, QD on Days 1-21, 840 mg IV of Atezo on Days 1 and 15, and 80 mg/m^2 IV Pac on Days 1, 8, and 15 of each 28-day cycle in expansion stage A3 until loss of clinical benefit, unacceptable toxicity, withdrawal of consent, or end of the study.
- Cohort 1- Arm C1: Participants with locally advanced or metastatic TNBC who had not previously received chemotherapy in the advanced setting received 400 mg of Ipat orally, QD on Days 1-21, 80 mg/m2 IV Pac on Days 1, 8, and 15 of Cycle 1 and 840 mg IV Atezo on Day 15 of Cycle 1 (1Cycle=28days). In Cycles ≥ 2, participants received 400 mg Ipat orally on Days 1-21, 840 mg IV Atezo on Days 1 and 15 and 80 mg/m2 IV Pac on Days 1, 8, and 15 of each 28-day Cycle during the safety run-in stage (C1) until loss of clinical benefit, unacceptable toxicity, withdrawal of consent, or end of the study.
- Cohort 1- Arm D2: Participants with locally advanced or metastatic TNBC received 840 mg IV Atezo on Days 1 and 15, 80 mg/m2 IV Pac on Days 1, 8, and 15 and 400 mg Ipat orally on days 15-21 of Cycle 1. In Cycles ≥ 2, participants received 400 mg Ipat orally on Days 1-21, 80 mg/m2 IV Pac on Days 1, 8, and 15 and 840 mg IV Atezo on Days 1 and 15 of each 28-day Cycle in the expansion stage D2 until loss of clinical benefit, unacceptable toxicity, withdrawal of consent, or end of the study.
Arm/Group | Cohort 1- Arm A1 | Cohort 1-Arm A2 | Cohort 1-Arm A3 | Cohort 1- Arm B1 | Cohort 1- Arm B2 | Cohort 1- Arm C1 | Cohort 1- Arm C2 | Cohort 1- Arm D1 | Cohort 1- Arm D2
Number analyzed (Participants) | 6 | 14 | 50 | 6 | 14 | 6 | 6 | 6 | 6
ng/mL
  Cycle 1 Day 15 Pre-dose: number analyzed (Participants) | 5 | 11 | 27 | 5 | 11 | 4 | 6 | 0 | 0
  Cycle 1 Day 15 Pre-dose | 27.0 (32.4) | 8.27 (404.3) | 15.0 (165.9) | 23.3 (58.3) | 24.1 (97.7) | 30.9 (48.3) | 36.4 (356.1) |  |
  Cycle 1 Day 15 1 hour Post-dose: number analyzed (Participants) | 5 | 10 | 25 | 5 | 10 | 0 | 0 | 0 | 0
  Cycle 1 Day 15 1 hour Post-dose | 200 (58.3) | 61.8 (209.2) | 85.9 (119.9) | 126 (158.4) | 86.4 (135.3) |  |  |  |
  Cycle 1 Day 15 2 hour Post-dose: number analyzed (Participants) | 5 | 10 | 33 | 5 | 10 | 0 | 0 | 6 | 4
  Cycle 1 Day 15 2 hour Post-dose | 151 (29.9) | 124 (55.0) | 153 (68.8) | 166 (102.2) | 120 (193.0) |  |  | 78.1 (125.6) | 177 (37.1)
  Cycle 1 Day 15 4 hour Post-dose: number analyzed (Participants) | 3 | 10 | 33 | 5 | 10 | 0 | 0 | 0 | 0
  Cycle 1 Day 15 4 hour Post-dose | 118 (26.1) | 121 (41.5) | 157 (62.9) | 154 (39.8) | 134 (99.2) |  |  |  |
  Cycle 1 Day 15 6 hour Post-dose: number analyzed (Participants) | 0 | 9 | 33 | 5 | 10 | 0 | 0 | 0 | 0
  Cycle 1 Day 15 6 hour Post-dose |  | 106 (47.3) | 133 (60.3) | 120 (45.6) | 101 (82.8) |  |  |  |
  Cycle 2 Day 15 Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 4 | 2
  Cycle 2 Day 15 Pre-dose |  |  |  |  |  | 22.5 (27.6) | 20.5 (38.4) | 15.2 (81.4) | 24.4 (76.7)
  Cycle 2 Day 15 1 hour Post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 4 | 2
  Cycle 2 Day 15 1 hour Post-dose |  |  |  |  |  | 41.3 (90.1) | 148 (39.4) | 70.5 (244.4) | 140 (94.2)
  Cycle 2 Day 15 2 hour Post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 4 | 2
  Cycle 2 Day 15 2 hour Post-dose |  |  |  |  |  | 206 (35.1) | 184 (28.0) | 120 (171.0) | 355 (22.9)
  Cycle 2 Day 15 4 hour Post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 3 | 2
  Cycle 2 Day 15 4 hour Post-dose |  |  |  |  |  | 185 (30.2) | 146 (46.5) | 131 (30.8) | 402 (43.4)
  Cycle 2 Day 15 6 hour Post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 5 | 3 | 2
  Cycle 2 Day 15 6 hour Post-dose |  |  |  |  |  | 124 (11.4) | 137 (30.4) | 98.8 (77.3) | 232 (57.4)
  Cycle 3 Day 15 1 to 3 hour Posst-dose: number analyzed (Participants) | 0 | 11 | 26 | 4 | 9 | 6 | 5 | 6 | 4
  Cycle 3 Day 15 1 to 3 hour Posst-dose |  | 47.1 (238.3) | 69.4 (161.2) | 68.6 (131.8) | 79.4 (150.8) | 50.4 (299.8) | 45.0 (182.3) | 84.6 (227.5) | 144 (121.6)

9. Secondary Outcome: Cohort 1 and Cohort 4: Number of Participants With Anti-Drug Antibodies (ADAs) for Atezolizumab During Study Treatment
Description: Participants were considered to be ADA positive if they were ADA negative or were missing data at Baseline but developed an ADA response following study drug exposure (treatment-induced ADA response), or if they were ADA positive at Baseline and the titer of one or more postbaseline samples was at least 0.60 titer unit greater than the titer of the Baseline sample (treatment-enhanced ADA response). Participants were considered to be ADA negative if they were ADA negative or had missing data at Baseline and all postbaseline samples were negative, or if they were ADA positive at Baseline but did not have any postbaseline samples with a titer that was at least 0.60 titer unit greater than the titer of the baseline sample (treatment unaffected). Since, Cohort 4 did not enroll any participants, data is only reported for Cohort 1.
Time Frame: From baseline up to 30 days from the last dose of atezolizumab (to approximately 4 years 1.1 month)
Population: Immunogenicity evaluable population included all participants with atleast 1 ADA assessment. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at a given time point.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1-Arm A1: Participants with locally advanced or metastatic TNBC who had not previously received chemotherapy in the advanced setting received 400 mg of Ipat orally, QD on Days 1-21, 840 mg IV of Atezo on Days 1 and 15, and 80 mg/m^2 IV Pac on Days 1, 8, and 15 of each 28-day cycle during the safety run-in stage (A1) until loss of clinical benefit, unacceptable toxicity, withdrawal of consent, or end of the study.
- Cohort 1- Arm A2: Participants with locally advanced or metastatic TNBC who had not previously received chemotherapy in the advanced setting received 400 mg of Ipat orally, QD on Days 1-21, 840 mg IV of Atezo on Days 1 and 15, and 80 mg/m^2 IV Pac on Days 1, 8, and 15 of each 28-day cycle in expansion stage A2 until loss of clinical benefit, unacceptable toxicity, withdrawal of consent, or end of the study.
- Cohort 1- Arm A3: Participants with locally advanced or metastatic TNBC who had not previously received chemotherapy in the advanced setting received 400 mg of Ipat orally, QD on Days 1-21, 840 mg IV of Atezo on Days 1 and 15, and 80 mg/m^2 IV Pac on Days 1, 8, and 15 of each 28-day cycle in expansion stage A3 until loss of clinical benefit, unacceptable toxicity, withdrawal of consent, or end of the study.
- Cohort 1-Arm B1: Participants with locally advanced or metastatic TNBC who had not previously received chemotherapy in the advanced setting received 400 mg of Ipat orally, QD on Days 1-21, 840 mg IV of Atezo on Days 1 and 15, and 100 mg/m^2 IV Nab-Pac on Days 1, 8, and 15 of each 28-day cycle during the safety run-in stage (B1) until loss of clinical benefit, unacceptable toxicity, withdrawal of consent, or end of the study.
- Cohort 1-Arm C1: Participants with locally advanced or metastatic TNBC who had not previously received chemotherapy in the advanced setting received 400 mg of Ipat orally, QD on Days 1-21, 80 mg/m2 IV Pac on Days 1, 8, and 15 of Cycle 1 and 840 mg IV Atezo on Day 15 of Cycle 1 (1Cycle=28days). In Cycles ≥ 2, participants received 400 mg Ipat orally on Days 1-21, 840 mg IV Atezo on Days 1 and 15 and 80 mg/m2 IV Pac on Days 1, 8, and 15 of each 28-day Cycle during the safety run-in stage (C1) until loss of clinical benefit, unacceptable toxicity, withdrawal of consent, or end of the study.
Arm/Group | Cohort 1-Arm A1 | Cohort 1- Arm A2 | Cohort 1- Arm A3 | Cohort 1-Arm B1 | Cohort 1- Arm B2 | Cohort 1-Arm C1 | Cohort 1- Arm C2 | Cohort 1- Arm D1 | Cohort 1- Arm D2
Number analyzed (Participants) | 6 | 13 | 43 | 6 | 14 | 6 | 6 | 6 | 6
Participants
  Baseline: Positive for ADA: number analyzed (Participants) | 6 | 13 | 43 | 6 | 14 | 0 | 0 | 6 | 6
  Baseline: Positive for ADA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline: Negative for ADA: number analyzed (Participants) | 6 | 13 | 43 | 6 | 14 | 0 | 0 | 6 | 6
  Baseline: Negative for ADA | 6 | 13 | 43 | 6 | 14 | 0 | 0 | 6 | 6
  Post Baseline: Positive for Treatment Emergent ADA: number analyzed (Participants) | 6 | 13 | 40 | 6 | 12 | 6 | 6 | 6 | 6
  Post Baseline: Positive for Treatment Emergent ADA | 0 | 3 | 2 | 0 | 3 | 2 | 1 | 0 | 0
  Post Baseline: Negative for Treatment Emergent ADA: number analyzed (Participants) | 6 | 13 | 40 | 6 | 12 | 6 | 6 | 6 | 6
  Post Baseline: Negative for Treatment Emergent ADA | 6 | 10 | 38 | 6 | 9 | 4 | 5 | 6 | 6

10. Secondary Outcome: Cohort 1 and Cohort 4: Plasma Concentration of Atezolizumab
Description: Since, Cohort 4 did not enroll any participants, data is only reported for Cohort 1.
Time Frame: Cycle 1 Day 1 and 15: predose and 30 mins post dose; Cycle 2: Day 1 and 15 predose, Cycle 3, 4, 8, 12, and 16 Day 1: predose; treatment discontinuation visit
Population: PK evaluable population included all participants who had at least 1 evaluable PK concentration post atezolizumab administration. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at a given time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Cohort 1-Arm C2: Participants with locally advanced or metastatic TNBC who had not previously received chemotherapy in the advanced setting received 400 mg of Ipat orally, QD on Days 1-21, 80 mg/m2 IV Pac on Days 1, 8, and 15 of Cycle 1 and 840 mg IV Atezo on Day 15 of Cycle 1 (1Cycle=28days). In Cycles ≥ 2, participants received 400 mg Ipat orally on Days 1-21, 840 mg IV Atezo on Days 1 and 15 and 80 mg/m2 IV Pac on Days 1, 8, and 15 of each 28-day Cycle in the expansion stage C2 until loss of clinical benefit, unacceptable toxicity, withdrawal of consent, or end of the study.
Arm/Group | Cohort 1- Arm A1 | Cohort 1-Arm A2 | Cohort 1-Arm A3 | Cohort 1- Arm B1 | Cohort 1- Arm B2 | Cohort 1-Arm C1 | Cohort 1-Arm C2 | Cohort 1- Arm D1 | Cohort 1- Arm D2
Number analyzed (Participants) | 6 | 14 | 50 | 6 | 14 | 6 | 6 | 6 | 6
ng/mL
  Cycle 1 Day 1 Pre-dose: number analyzed (Participants) | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 2 | 0
  Cycle 1 Day 1 Pre-dose |  |  | 853 (1344.8) |  | 65.3 (3.4) |  |  | 82.5 (7.6) |
  Cycle 1 Day 1 30 min Post-dose: number analyzed (Participants) | 4 | 13 | 37 | 5 | 12 | 0 | 0 | 6 | 5
  Cycle 1 Day 1 30 min Post-dose | 354000 (12.2) | 330000 (18.1) | 329000 (25.3) | 315000 (5.4) | 365000 (19.2) |  |  | 335000 (13.9) | 339000 (13.6)
  Cycle 1 Day 15 Pre-Dose: number analyzed (Participants) | 5 | 10 | 40 | 5 | 11 | 1 | 0 | 5 | 5
  Cycle 1 Day 15 Pre-Dose | 106000 (12.1) | 75200 (170.2) | 94500 (27.8) | 93100 (15.6) | 91700 (21) | 126 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. |  | 87100 (31.6) | 108000 (32.2)
  Cycle 1 Day 15 30 min Post-dose: number analyzed (Participants) | 0 | 0 | 14 | 0 | 1 | 4 | 4 | 1 | 1
  Cycle 1 Day 15 30 min Post-dose |  |  | 351000 (49) |  | 393000 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 362000 (8.8) | 370000 (9.8) | 274000 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 345000 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated.
  Cycle 2 Day 1 Pre-Dose: number analyzed (Participants) | 5 | 11 | 33 | 6 | 12 | 5 | 6 | 6 | 6
  Cycle 2 Day 1 Pre-Dose | 143000 (34.3) | 90200 (883.4) | 149000 (45) | 99700 (118.4) | 132000 (45) | 101000 (39.1) | 121000 (21.6) | 147000 (35.3) | 156000 (20)
  Cycle 2 Day 15 Pre-Dose: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 5 | 4 | 3 | 2
  Cycle 2 Day 15 Pre-Dose |  |  | 120000 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. |  | 180000 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 124000 (83.8) | 189000 (18.2) | 178000 (41.7) | 194000 (26.1)
  Cycle 3 Day 1 Pre-Dose: number analyzed (Participants) | 6 | 12 | 30 | 6 | 11 | 5 | 5 | 5 | 4
  Cycle 3 Day 1 Pre-Dose | 193000 (85.5) | 105000 (1195.9) | 216000 (50.7) | 219000 (32) | 246000 (33) | 166000 (34.7) | 230000 (16.1) | 197000 (32.4) | 247000 (9.7)
  Cycle 4 Day 1 Pre-Dose: number analyzed (Participants) | 5 | 11 | 22 | 6 | 10 | 6 | 5 | 6 | 4
  Cycle 4 Day 1 Pre-Dose | 347000 (12.4) | 179000 (256.2) | 283000 (23.8) | 239000 (37) | 283000 (16.7) | 293000 (40.3) | 293000 (18.3) | 250000 (43.9) | 247000 (46)
  Cycle 8 Day 1 Pre-Dose: number analyzed (Participants) | 5 | 6 | 6 | 3 | 4 | 4 | 2 | 3 | 2
  Cycle 8 Day 1 Pre-Dose | 376000 (11.9) | 398000 (34.4) | 345000 (55.9) | 385000 (19.2) | 293000 (7.1) | 386000 (32.5) | 545000 (29.6) | 153000 (119.9) | 357000 (10.3)
  Cycle 12 Day 1 Pre-Dose: number analyzed (Participants) | 1 | 3 | 0 | 0 | 1 | 1 | 2 | 2 | 0
  Cycle 12 Day 1 Pre-Dose | 333000 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 505000 (14.4) |  |  | 285000 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 122000 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 384000 (11.8) | 393000 (26) |
  Cycle 16 Day 1Pre-Dose: number analyzed (Participants) | 3 | 5 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Cycle 16 Day 1Pre-Dose | 562000 (40.3) | 408000 (42) |  | 388000 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. |  | 135000 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. |  |  |
  Treatment Discontinuation: number analyzed (Participants) | 0 | 5 | 8 | 4 | 8 | 2 | 2 | 3 | 3
  Treatment Discontinuation |  | 97400 (153.2) | 135000 (99.8) | 253000 (81.9) | 195000 (47.5) | 337000 (31.7) | 181000 (40.9) | 274000 (113) | 178000 (67.9)

11. Secondary Outcome: Cohort 1 and Cohort 4: Clinical Benefit Rate (CBR) as Assessed by Investigator Based on RECIST v1.1
Description: CBR was defined as percentage of participants with stable disease (SD) for at least 24 weeks or with confirmed CR or PR as determined by the investigator according to RECIST v1.1. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum on study. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. Since, Cohort 4 did not enroll any participants, data is only reported for Cohort 1.
Time Frame: From screening up to confirmed SD or CR or PR (up to approximately 43.6 months)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1-Arm A | Cohort 1-Arm B | Cohort 1-Arm C | Cohort 1-Arm D
Number analyzed (Participants) | 70 | 20 | 12 | 12
percentage of participants | 58.6 [46.17 to 70.23] | 65.0 [40.78 to 84.61] | 75.0 [42.81 to 94.51] | 58.3 [27.67 to 84.83]

ADVERSE EVENTS:
Time Frame: Up until 90 days after the last dose of study treatment or until initiation of new systemic anti-cancer therapy, whichever occurs first (up to 4 years 1 month)
Description: Safety population included all participants who received any study treatment. No participants enrolled in Arm G and H, and hence no data was reported.
Groups:
- Cohort 1- Arm A: Participants with locally advanced or metastatic triple-negative breast cancer (TNBC) who had not previously received chemotherapy in the advanced setting received 400 milligrams (mg) of ipatasertib (Ipat) orally, once daily (QD) on Days 1-21, 840 mg intravenous (IV) of atezolizumab (Atezo) on Days 1 and 15, and 80 milligrams per square meter (mg/m^2) IV paclitaxel (Pac) on Days 1, 8, and 15 of each 28-day cycle. Following completion of a safety run-in cohort (A1), subsequent expansion arms enrolled (A2 and A3). All participants in Arm A continued to receive treatment until loss of clinical benefit, unacceptable toxicity, withdrawal of consent, or end of the study.
- Cohort 1- Arm B: Participants with locally advanced or metastatic TNBC who had not previously received chemotherapy in the advanced setting received 400 mg of Ipat orally, QD on Days 1-21, 840 mg IV of Atezo on Days 1 and 15, and 100 mg/m^2 IV nab-paclitaxel (Nab-Pac) on Days 1, 8, and 15 of each 28-day cycle. Following completion of a safety run-in cohort (B1), a subsequent expansion arm enrolled (B2). All participants in Arm B continued to receive treatment until loss of clinical benefit, unacceptable toxicity, withdrawal of consent, or end of the study.
- Cohort 1- Arm C: Participants with locally advanced or metastatic TNBC who had not previously received chemotherapy in the advanced setting received 400 mg of Ipat orally, QD on Days 1-21, 80 mg/m2 IV Pac on Days 1, 8, and 15 and 840 mg IV Atezo on Day 15 of Cycle 1 (28 day cycle). In Cycles ≥ 2, participants received 400 mg Ipat orally on Days 1-21, 840 mg IV Atezo on Days 1 and 15 and 80 mg/m2 IV Pac on Days 1, 8, and 15 of each 28-day Cycle. Following completion of the safety run-in cohort (C1), a subsequent expansion cohort (C2) enrolled. All participants in Arm C continued to receive treatment until loss of clinical benefit, unacceptable toxicity, withdrawal of consent, or end of the study.
- Cohort 1- Arm D: Participants with locally advanced or metastatic TNBC who had not previously received chemotherapy in the advanced setting received 840 mg IV Atezo on Days 1 and 15, 80 mg/m2 IV Pac on Days 1, 8, and 15 and 400 mg Ipat orally on days 15-21 of Cycle 1 (28 day cycle). In Cycles ≥ 2, participants received 400 mg Ipat orally on Days 1-21, 80 mg/m2 IV Pac on Days 1, 8, and 15 and 840 mg IV Atezo on Days 1 and 15 of each 28 day Cycle. Following completion of the safety run-in cohort (D1), a subsequent expansion cohort (D2) enrolled. All participants in Arm D continued to receive treatment until loss of clinical benefit, unacceptable toxicity, withdrawal of consent, or end of the study.
- Cohort 2- Arm E: Participants in the second-line and third-line setting with locally advanced or metastatic TNBC received 400 mg Ipat orally QD on Days 1-28 and 840 mg IV Atezo on Days 8 and 22 of Cycle 1 (Cycle 1 = 35 days). In Cycles ≥ 2, participants received 400 mg Ipat orally on Days 1-21 and 840 mg IV Atezo on Days 1 and 15 of each cycle (Cycles ≥ 2 = 28 days) until loss of clinical benefit, unacceptable toxicity, withdrawal of consent, or end of the study.
- Cohort 3- Arm F: Participants in the safety run-in stage (arm F1) with locally advanced T2-4 TNBC received 300 mg Ipat orally QD on Days 1-21, 840mg IV Atezo on Days 1 and 15, 60 mg/m2 IV doxorubicin and 600 mg/m2 IV cyclophosphamide on Days 1 and 15 of Cycles 1 and 2 (1 Cycle=28-days). Participants then received 400 mg Ipat orally QD on Days 1-21, 840mg IV Atezo on Days 1 and 15 and 80 mg/m2 IV Pac on Days 1, 8, 15, and 22 of Cycles 3-5, until completion of 5 cycles or disease progression or unacceptable toxicity, whichever occurred first.
Arm/Group | Cohort 1- Arm A | Cohort 1- Arm B | Cohort 1- Arm C | Cohort 1- Arm D | Cohort 2- Arm E | Cohort 3- Arm F
All-Cause Mortality (participants affected / at risk) | 34/70 | 16/20 | 5/12 | 5/12 | 10/17 | 0/6
Serious Adverse Events (participants affected / at risk) | 26/70 | 9/20 | 5/12 | 4/12 | 5/17 | 4/6
Other Adverse Events (participants affected / at risk) | 70/70 | 20/20 | 12/12 | 12/12 | 17/17 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1- Arm A (N=70) | Cohort 1- Arm B (N=20) | Cohort 1- Arm C (N=12) | Cohort 1- Arm D (N=12) | Cohort 2- Arm E (N=17) | Cohort 3- Arm F (N=6)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin I increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperamylasaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1- Arm A (N=70) | Cohort 1- Arm B (N=20) | Cohort 1- Arm C (N=12) | Cohort 1- Arm D (N=12) | Cohort 2- Arm E (N=17) | Cohort 3- Arm F (N=6)
Anaemia (Blood and lymphatic system disorders) | 17 (20) | 6 (10) | 3 (5) | 2 (3) | 1 (1) | 4 (5)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 15 (43) | 3 (6) | 2 (6) | 2 (5) | 1 (1) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 5 (6) | 1 (1) | 2 (2) | 3 (5) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 7 (8) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Xerophthalmia (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 12 (15) | 2 (2) | 3 (3) | 3 (4) | 0 (0) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 5 (6) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 25 (34) | 7 (8) | 4 (6) | 5 (6) | 3 (3) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 59 (127) | 15 (51) | 10 (22) | 9 (18) | 9 (14) | 6 (19)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 10 (11) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 37 (55) | 16 (29) | 4 (4) | 5 (10) | 5 (7) | 5 (9)
Stomatitis (Gastrointestinal disorders) | 8 (12) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 15 (29) | 11 (19) | 4 (5) | 3 (3) | 3 (3) | 1 (1)
Asthenia (General disorders) | 19 (28) | 7 (12) | 3 (3) | 4 (9) | 9 (10) | 3 (6)
Chest pain (General disorders) | 3 (3) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 32 (46) | 6 (8) | 5 (9) | 4 (5) | 2 (2) | 2 (2)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 2 (3) | 2 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 5 (7) | 1 (3) | 1 (1) | 2 (3) | 2 (3) | 1 (2)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 5 (7) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 17 (26) | 6 (6) | 5 (12) | 1 (3) | 4 (4) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alveolar osteitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Genital herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 3 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 7 (9) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 8 (9) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular access site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 10 (15) | 0 (0) | 1 (1) | 3 (6) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular access site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 14 (22) | 2 (2) | 1 (4) | 3 (7) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 4 (4) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 9 (13) | 1 (1) | 2 (7) | 3 (6) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Blood creatinine increased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 3 (5) | 1 (2) | 2 (3) | 2 (7) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (5) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 2 (3) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 14 (17) | 3 (4) | 1 (1) | 4 (4) | 3 (3) | 1 (1)
Food intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (6) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (8) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (15) | 2 (5) | 4 (4) | 2 (2) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (14) | 4 (5) | 3 (4) | 1 (1) | 0 (0) | 2 (2)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (9) | 1 (1) | 2 (3) | 2 (2) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (9) | 1 (1) | 2 (3) | 1 (1) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 6 (7) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dysaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 8 (9) | 2 (2) | 1 (2) | 2 (2) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 19 (29) | 4 (4) | 2 (2) | 1 (1) | 5 (6) | 1 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 20 (24) | 9 (11) | 7 (8) | 0 (0) | 1 (1) | 0 (0)
Neurotoxicity (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Paraesthesia (Nervous system disorders) | 9 (9) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (7) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sensory disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (4) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Euphoric mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 5 (6) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 3 (4) | 2 (3) | 2 (2) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 26 (27) | 11 (13) | 6 (6) | 7 (7) | 0 (0) | 4 (4)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 5 (7) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (7) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Onychalgia (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prurigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (15) | 4 (4) | 3 (4) | 2 (2) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 25 (39) | 8 (11) | 3 (14) | 4 (4) | 7 (7) | 3 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 4 (4) | 3 (3) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 5 (5) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ocular discomfort (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papilloedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Animal scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cortisol decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema annulare (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-26): https://cdn.clinicaltrials.gov/large-docs/36/NCT03800836/Prot_SAP_000.pdf